CLINICAL TRIAL: NCT05488275
Title: Prospective, Randomized, Double Blinded Trial Comparing Medial Patellofemoral Ligament Reconstruction (Hamstrings) Versus Campbell Functional Reconstruction (Non-anatomic) in Recurrent Patella Dislocation
Brief Title: MPFL vs Campbell in Recurrent Patella Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Clinical Professor, Head of Knee Surgery Division and Arthroscopy, Department of Trauma Surgery and Orthopedics, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: mpfl_campbell
Record Dates: First submitted 2020-07-18; First posted 2022-08-04 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Patella Dislocation
Keywords: MPFL; Campbell
MeSH Terms: conditions — Patellar Dislocation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MPFL static (Active Comparator): Medial Patellofemoral Ligament reconstruction with hamstring graft - static procedure
  Interventions: Procedure: Surgery
- Campbell (Active Comparator): Medial Patellofemoral Ligament reconstruction using non-anatomic reconstruction (quadriceps femoris plasty - Campbell method)
  Interventions: Procedure: Surgery
- MPFL dynamic (Active Comparator): Medial Patellofemoral Ligament reconstruction with hamstring graft - dynamic procedure
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — MPFL reconstruction

SUMMARY:
This study will compare anatomic Medial Patellofemoral Reconstruction from Hamstring graft with non anatomic reconstruction according to Campbell. The purpose of this study is to evaluate which type of treatment recurrent patella dislocation provides to better clinical, radiological and laboratory outcomes.

DETAILED DESCRIPTION:
Recurrent patella dislocation require surgery treatment. It provides to less cartilage degeneration and slow down knee osteoarthritis. Medial retinacular complex is injured in first time patella dislocation and its reconstruction is necessary. In literature there can be found many surgical reconstruction technics: anatomical or non anatomical (functional). But there is lack of evidence which technic provides to better outcomes - reduce the possibility to patella dislocation and progression of osteoarthritis in patellofemoral joint. Nowadays the choice of performed surgery depends on surgeons personal assessment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent patella dislocation
* No patellofemoral joint dysplasia or Dysplasia A/B according to Dejour (non operating)
* Acceptable is to perform concomitant medialization Tibial Tubercle Osteotomy

Exclusion Criteria:

* no informed consent to participate in the study
* age under 18 years or above 65
* multiligament injury or single plane knee instability
* another musculoskeletal disorders in lower limb
* lower limb deformity requiring axis correction: valgus
* femoral anteversion (CT measurements)
* joints inflammatory diseases
* concomitant patellectomy or trochleoplasty
* ASA score > II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Imaging modality X-ray | 1 year
  Patellofemoral Joints Biomechanics improvement measured by patella tilt
Imaging modality X-ray | 2 years
  Patellofemoral Joints Biomechanics improvement measured by Q angle
Imaging modality CT | 2 years
  Patellofemoral Joints Biomechanics improvement measured by Insall-Salvati ratio. The Insall-Salvati ratio or index is the ratio of the patella tendon length to the length of the patella and is used to determine patellar height. he Insall-Salvati ratio was initially determined on a 30° flexed lateral knee x-ray and was later applied to sagittal MRI.
  Distance lines are used to calculate Insall-Salvati ratio:
  A: patellar tendon length (TL): length of the posterior surface of the tendon from the lower pole of the patella to its insertion on the tibia B: patellar length (PL): greatest pole-to-pole length Insall-Salvati ratio = A/B (or TL/PL). patella baja: <0.8 normal: 0.8-1.2 patella alta: >1.2
Imaging modality CT | 2 years
  Patellofemoral Joints Biomechanics improvement measured by TT-TG (line between tibial tuberosity and trochlear groove)

SECONDARY OUTCOMES:
Functional tests | 12 weeks
  hop-for-distance
Functional tests | 6 months
  hop-for-distance
Functional tests | 12 months
  hop-for-distance
Functional tests | 24 months
  hop-for-distance
Knee Injury and Osteoarthritis Outcome Score | 12 weeks,
  Knee Injury and Osteoarthritis Outcome Score; The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee Injury and Osteoarthritis Outcome Score | 6 months,
  Knee Injury and Osteoarthritis Outcome Score;The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems. KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee Injury and Osteoarthritis Outcome Score | 12 months
  Knee Injury and Osteoarthritis Outcome Score; The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee Injury and Osteoarthritis Outcome Score | 24 months
  Knee Injury and Osteoarthritis Outcome Score;The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems. KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
International Knee Documentation Committee | 12 weeks
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. higher number representing higher levels of function.
International Knee Documentation Committee | 6 months
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. higher number representing higher levels of function.
International Knee Documentation Committee | 12 months
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. higher number representing higher levels of function.
International Knee Documentation Committee | 24 months
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. higher number representing higher levels of function.
Tegner Lysholm Knee Scoring Scale | 12 weeks,
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 6 months,
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 12 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Pain Visual Analog Scale | 12 weeks,
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Pain Visual Analog Scale | 6 months,
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Pain Visual Analog Scale. | 12 months,
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Pain Visual Analog Scale | 24 months
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Knee Injury and Osteoarthritis Outcome Score Patellofemoral | 12 weeks
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
Knee Injury and Osteoarthritis Outcome Score Patellofemoral | 6 months,
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
Knee Injury and Osteoarthritis Outcome Score Patellofemoral | 12 months
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
Knee Injury and Osteoarthritis Outcome Score Patellofemoral | 24 months
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
The Victorian Institute of Sport Assessment | 12 weeks,
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. minimum 0, maximum 100 for asymptomatic
The Victorian Institute of Sport Assessment | 6 months,
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. minimum 0, maximum 100 for asymptomatic
The Victorian Institute of Sport Assessment | 12 months,
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. minimum 0, maximum 100 for asymptomatic
The Victorian Institute of Sport Assessment | 24 months
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. minimum 0, maximum 100 for asymptomatic

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kamiński, Principal Investigator — PCME, Otwock, Poland
Locations (1):
- Department of Orthopaedics and Traumatology, Postgraduate Center for Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland